CLINICAL TRIAL: NCT03864991
Title: Lifestyle Changes and Glycemic Control in Type 1 Diabetes Mellitus: A Factorial Design Approach
Brief Title: Lifestyle Changes and Glycemic Control in T1D
Acronym: LSHBA1C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Syed Iqbal Azam, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 5363-CHS-ERC-18
Record Dates: First submitted 2019-02-28; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Type1 Diabetes Mellitus; Life Style; Behavioral Changes; Self-Management
Keywords: Log book; Step count; Diet; Physical activity; HbA1c; Blood sugar
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A factorial design approach will be taken to study the lifestyle change for self-management of T1D. A randomized controlled method will enroll patients in four groups. All groups will be working with a standard log book for documenting blood sugar and routine care as advise by doctors, nurses, and nutritionists. First group will be entirely of routine care follow up, second group will receive additional e-device for step count (fitbit), third group will receive routine care and e-messages as reminders to maintain a daily log book, and fourth group will be receiving e-device for step count (fitbit) and e-messages for maintain blood glucose and step count log book in addition to routine care. All four groups will be followed up for a period of six months. Log book data will be obtained at a monthly interval and HbA1c as a main outcome will be measured three times, at baseline, at three and six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Routine Care (No Intervention): This group will be followed up for routine care, maintaining a standard log book for documenting blood sugar and insulin dosages per advice and explanation by doctors, nurses and nutritionists.
- e-device for step count (fit-bit) (Active Comparator): This group will receive e-device for step count (fit-bit) in addition to routine care.
  Interventions: Device: e-device for step count (fit-bit)
- e-messages for log book (Active Comparator): This group will receive daily e-messages for maintaining log book in addition to routine care.
  Interventions: Behavioral: e-messages for log book
- e-messages for log book & fit-bit (Active Comparator): This group will receive e-device for step count (fit-bit), daily e-messages for maintaining log book for blood sugar, insulin dosages and step count in addition to routine care.
  Interventions: Device: e-device for step count (fit-bit); Behavioral: e-messages for log book & fit-bit

INTERVENTIONS:
Device: e-device for step count (fit-bit) — Patients in this group will receive fitbit device to count their daily steps and record it into their log books.
  Arms: e-device for step count (fit-bit); e-messages for log book & fit-bit
Behavioral: e-messages for log book — Patients in this group will receive e-messages to maintain their log books as per instruction for blood sugar levels and send back weekly through snap shot.
  Arms: e-messages for log book
Behavioral: e-messages for log book & fit-bit — Patient in this group will receive e-messages to maintain their log books for blood sugar levels as well as use fitbit device and maintain their log book for daily step count and send back weekly through snap shot.
  Arms: e-messages for log book & fit-bit

SUMMARY:
Pakistani studies report non-adherence to self-management by type 1 diabetes (T1D) patients, and episodes of hypoglycemia and ketoacidosis as acute complications. Self-management guidelines include maintenance of logbooks for blood glucose, physical activity, and dietary intake, that affect glycated hemoglobin (HbA1C) and acute complications. The proposed study will evaluate whether mobile messaging for maintaining log books for blood glucose or e-device use for step count will modify HbA1c levels to be examined at three and six months after enrollment. In addition, episodes of acute complications and blood glucose variability will be correlated with daily log book maintenance and step counts.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) occurs due to destruction of insulin producing beta cells in pancreas. T1D usually occurs in children and young individuals, and requires continuous blood glucose monitoring for adjustment of insulin dosage on a daily basis. Incidence of T1D has been increasing over the past three decades. Hyperglycemia and ketoacidosis episodes are common adverse effects due to irregular monitoring of daily blood glucose. It is a big challenge in developed as well as developing countries to live with T1D due to less optimal use of timely entry in logbook for self-monitoring of blood glucose (SMBG). Current guidelines recommend SMBG use in all patients with diabetes. According to a study, increased daily frequency of SMBG was significantly associated with lower glycated hemoglobin (HbA1C) along with added benefits of fewer acute complications among children and adolescents. Available literature from Pakistan highlights non-adherence of T1D patients to recommended dietary advice (58.5%), physical activity (42.3%) and prescribed insulin regimen (88.1%). Use of mobile applications has been shown to increase the medication adherence and use of self-blood glucose testing. Increased daily step count by T1D patients helped to reduce the risk of cardiovascular events. A wearable e-device accompanied with an application (Fitbit App) tracks step count by recording data in mobile application. HbA1C levels acts as an indicator for the glycemic control and correlates with complications. However, HbA1C cannot determine the daily variability of blood glucose, thus SMBG can help predict the average daily risk reduction in T1D complications. The proposed study will address the adherence to standard protocols for maintaining home based records by patients and caregivers and insulin therapy, optimizing the quarterly HbA1C levels.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with T1D > 6 months
* Patient's age ≥ 15 years
* Patient or any one of the family member like father, mother or sibling using smart phone.
* Patient or any one of the family member know how to use (receive calls or read text message) a smart phone.

Exclusion Criteria:

* Patient on insulin pump
* Pregnant females,
* Patient with neurodevelopmental delay or thalassemia
* Patient currently using any kind of authentic e-device for step count or physical activity.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1c | Each participant will be in the study for the period of six months
  Blood HbA1c levels will be measured at baseline, three and six months. It will be taken on ratio scale measured in mmol/mol

SECONDARY OUTCOMES:
Episodes of acute complications | Each participant will be in the study for the period of six months
  Hyperglycemia >450 mg/dl or "Hi" on glucometer, Ketoacidosis per hospital diagnosed, Hypoglycemia <60 mg/dl or "low" on glucometer three times a day.

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Azam, MSc, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sawani S, Siddiqui AR, Azam SI, Humayun K, Ahmed A, Habib A, Naz S, Tufail M, Iqbal R. Lifestyle changes and glycemic control in type 1 diabetes mellitus: a trial protocol with factorial design approach. Trials. 2020 Apr 20;21(1):346. doi: 10.1186/s13063-020-4205-7. PMID 32312302